CLINICAL TRIAL: NCT05850403
Title: Social Media Impact on Patients' Decision-Making Regarding Aesthetic Dental Treatments: A Web-Based Questionnaire Study
Brief Title: Social Media Impact on Patients' Regarding Aesthetic Dental Treatments
Status: Completed | Type: Observational
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Freire Mancebo, Principal Investigator, Universidad Europea de Madrid
Other Study IDs: 22.022
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Social Media; Dentist-Patient Relations
Keywords: Social Media; Dentist-Patient Relations; Aesthetic dentistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study was to describe dental patients the use of social media related to aesthetic dental treatments. The main questions it aims to answer were:

* Describe the use of social media before undergoing an aesthetic treatment.
* To assess the influence of social media prior to undergoing aesthetic treatment

Participants answered a web-base questionnaire.

DETAILED DESCRIPTION:
In recent years, an increased use of social media has been observed. Therefore, the aim of this observational study is to describe the use of social media in dental patients in relation to aesthetic dental treatments, as well as, its possible influence. A 25-question questionnaire was designed with the following 4 sections: (i) informed consent; (ii) demographic characteristics; (iii) cosmetic dental treatments; and (iv) social media use.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old that use social media

Exclusion Criteria:

* Not having undergone any aesthetic dental treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Undergraduate students meeting the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Use of social media | 3 minutes
  Percentage of participants that used social media when undergoing aesthetic dental treatment

SECONDARY OUTCOMES:
Influence of social media | 3 minutes
  Percentage of participants that social media influenced them when undergoing aesthetic dental treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No